CLINICAL TRIAL: NCT00039377
Title: A Phase II Trial of Sequential Chemotherapy, Imatinib Mesylate (Gleevec, STI571) (NSC # 716051), and Transplantation for Adults With Newly Diagnosed Ph+ Acute Lymphoblastic Leukemia by the CALGB and SWOG
Brief Title: Chemotherapy, Imatinib Mesylate, and Peripheral Stem Cell Transplantation in Treating Patients With Newly Diagnosed Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00436; NCI-2009-00436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000069378; CALGB 10001/SWOG C10001 (Other: Cancer and Leukemia Group B); CALGB-10001 (Other: CTEP); U10CA031946 (NIH); NCT01648426 (obsolete NCT alias)
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Results first posted 2014-03-18 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-06

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission
MeSH Terms: interventions — Imatinib Mesylate; Methotrexate; merphos; Vincristine; Leucovorin; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation; Tacrolimus; Filgrastim; Granulocyte Colony-Stimulating Factor; Etoposide; Cyclophosphamide; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (imatinib mesylate, chemotherapy, PBSCT) (Experimental): See Detailed Description.
  Interventions: Drug: imatinib mesylate; Drug: methotrexate; Drug: vincristine sulfate; Drug: leucovorin calcium; Procedure: peripheral blood stem cell transplantation; Procedure: autologous hematopoietic stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Radiation: total-body irradiation; Drug: tacrolimus; Biological: filgrastim; Drug: etoposide; Drug: cyclophosphamide; Drug: cytarabine; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: imatinib mesylate — Given PO
  Other Names: CGP 57148; Gleevec; Glivec
Drug: methotrexate — Given IT and IV
  Other Names: amethopterin; Folex; methylaminopterin; Mexate; MTX
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: leucovorin calcium — Given IV and PO
  Other Names: CF; CFR; LV
Procedure: peripheral blood stem cell transplantation — Undergo PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: autologous hematopoietic stem cell transplantation — Undergo autologous PBSCT
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo allogeneic PBSCT
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: tacrolimus — Given IV or PO
  Other Names: FK 506; Prograf
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial studies how well giving imatinib mesylate together with chemotherapy and peripheral stem cell transplantation works in treating patients with newly diagnosed acute lymphoblastic leukemia. Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Imatinib mesylate may stop the growth of cancer cells by blocking the enzymes necessary for cancer cell growth. Giving imatinib mesylate together with chemotherapy and peripheral stem cell transplantation may be an effective treatment for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the activity of imatinib mesylate (Gleevec) to prolong disease-free survival (DFS) and overall survival in acute lymphoblastic leukemia (ALL) patients with t(9;22).

II. Determine the ability of imatinib mesylate (Gleevec) to produce or maintain a BCR-ABL-negative status, as judged by real-time-polymerase chain reaction (RT-PCR) following sequential chemotherapy, imatinib mesylate (Gleevec) and transplantation.

III. Determine the feasibility of collecting adequate peripheral blood stem cells for autologous transplantation following imatinib mesylate (Gleevec) therapy.

IV. Study the safety and efficacy of autologous peripheral stem cell transplantation following therapy with imatinib mesylate (Gleevec).

V. Study the safety and efficacy of allogeneic stem cell transplantation following therapy with imatinib mesylate (Gleevec).

VI. Study the safety and efficacy of imatinib mesylate (Gleevec) administered after allogeneic or autologous stem cell transplant.

OUTLINE:

COURSE I (remission induction): Patients receive 1 course of front-line induction therapy on a Cancer and Leukemia Group B (CALGB)/Southwest Oncology Group (SWOG) protocol prior to enrollment.

COURSE II (imatinib mesylate): Patients receive imatinib mesylate orally (PO) twice daily on days 1-28.

COURSE III (CNS prophylaxis): Within 7 days after completing course II, patients receive methotrexate intrathecally (IT), methotrexate intravenously (IV) over 3 hours, and vincristine sulfate IV on days 1, 8, and 15; methotrexate PO every 6 hours on days 1-2, 8-9, and 15-16; leucovorin calcium IV on days 2, 9, and 16; and leucovorin calcium PO every 6 hours on days 3, 4, 10, 11, 17, and 18.

COURSE IV (imatinib mesylate): After blood counts recover after completion of course III, patients receive imatinib mesylate as in course II.

COURSE V: Patients undergo allogeneic peripheral blood stem cell transplantation (PBSCT), autologous PBSCT, or no PBSCT.

COURSE Va (allogeneic PBSCT for patients with human leukocyte antigen [HLA]-matched sibling donor): Beginning 3-10 days after completion of course IV, patients with an HLA-matched sibling donor undergo total body irradiation (TBI) 2-3 times daily on days -7 to -4. Patients receive etoposide IV over 4 hours on day -3. Patients then undergo PBSCT on day 0. Patients then receive graft-vs-host disease prophylaxis with tacrolimus IV continuously on days -1 to 56 (or IV continuously on days -1 to 14 and then PO or IV every 12 hours on days 15-56) followed by a taper. Patients also receive methotrexate IV on days 1, 3, and 6, and filgrastim subcutaneously (SC) beginning on day 4 and continuing until blood counts recover.

COURSE Vb (autologous PBSCT for patients without HLA-matched sibling donor): Beginning 3-10 days after completion of course IV, patients without an HLA-matched sibling donor receive etoposide IV continuously and cytarabine IV over 2 hours on days 1-4. Patients also receive filgrastim SC beginning on day 14 and continuing until PBSC collection is complete. Patients receive imatinib mesylate PO twice daily beginning after completion of PBSC collection and continuing until 3 days before PBSCT. Patients then undergo TBI 2-3 times daily on days -8 to -5. Patients receive etoposide IV over 4 hours on day -4 and cyclophosphamide IV over 2 hours on day -2. Patients undergo PBSCT on day 0. Patients receive filgrastim SC beginning on day 0 and continuing until blood counts recover.

COURSE Vc (no transplantation for patients who are not transplant candidates): Beginning 3-10 days after completion of course IV, patients who are not candidates for PBSCT receive etoposide IV over 4 hours and cytarabine IV over 2 hours on days 1-4. Patients also receive filgrastim SC once or twice a day beginning on day 14 and continuing until blood counts recover.

COURSE VI: Patients receive imatinib mesylate PO once or twice daily beginning on day 30 post transplantation or on day 30 if no transplantation received and continuing for at least 1 year or until patient has 2 consecutive negative reverse transcriptase-polymerase chain reaction assays at least 3 months apart or until relapse.

After completion of study treatment, patients are followed up monthly for 1 year, every 3 months for 2 years, every 6 months for 2 years, then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologic diagnosis of ALL
* Detection of the t(9;22)(q34;q11) or 3-way variant by metaphase cytogenetics or BCR-ABL positive by molecular analysis (RT-PCR or fluorescence in situ hybridization [FISH})
* Prior Therapy:

  * Complete or partial remission following one course of induction chemotherapy with an intensive 4 or 5 drug regimen (with or without imatinib mesylate) on a CALGB or SWOG ALL protocol for previously untreated ALL patients

    * Note: The double induction regimen of SWOG S0333 is considered to be one course of induction chemotherapy for the purpose of this eligibility criterion; therefore, patients from S0333 may be eligible for this study only after completing the entire double induction regimen
  * Complete or partial remission following one course of therapy on any standard induction regimen (with or without imatinib mesylate) without prior enrollment on a cooperative group frontline protocol; in these instances, documentation of Philadelphia chromosome (Ph)+ positivity may occur outside a CALGB or SWOG laboratory

    * Note: CALGB institutions must enroll patients on CALGB 9862 and submission of an initial sample for the companion trial must occur at time of enrollment on CALGB C10001; enrollment on companion studies CALGB 8461 and 9665 is not required
* No more than six weeks of prior imatinib mesylate during induction therapy before study enrollment
* Non-pregnant and non-nursing; treatment under this protocol would expose an unborn child to significant risks; women and men of reproductive potential should agree to use an effective means of birth control and contraception should continue for three months after the last dose of imatinib mesylate (Gleevec) to allow complete clearance of drug and its principle metabolites from the body; in women of childbearing potential, a pregnancy test will be required at study entry

Ages: 15 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 58 (Actual)
Dates: Start 2002-04; Primary Completion 2012-04 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meir Wetzler, Principal Investigator — Cancer and Leukemia Group B
Locations (97):
- United States (97):
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - University of Chicago, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Eureka Hospital, Eureka, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Radiation Oncology Center of Olathe, Olathe, Kansas
  - Radiation Oncology Practice Corporation Southwest, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Eastern Maine Medical Center, Bangor, Maine
  - Beverly Hospital, Beverly, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Commonwealth Hematology Oncology PC-Worcester, Worcester, Massachusetts
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Radiation Oncology Practice Corporation South, Kansas City, Missouri
  - Radiation Oncology Practice Corporation - North, Kansas City, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine of Bozeman, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Frisbie Hospital, Rochester, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Manhasset, New York
  - North Shore-LIJ Health System CCOP, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - North Shore-LIJ Health System/Center for Advanced Medicine, New Hyde Park, New York
  - Weill Medical College of Cornell University, New York, New York
  - Oswego Hospital, Oswego, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Northeastern, St. Johnsbury, Vermont
  - Virginia Commonwealth University, Richmond, Virginia
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Wetzler M, Watson D, Stock W, Koval G, Mulkey FA, Hoke EE, McCarty JM, Blum WG, Powell BL, Marcucci G, Bloomfield CD, Linker CA, Larson RA. Autologous transplantation for Philadelphia chromosome-positive acute lymphoblastic leukemia achieves outcomes similar to allogeneic transplantation: results of CALGB Study 10001 (Alliance). Haematologica. 2014 Jan;99(1):111-5. doi: 10.3324/haematol.2013.085811. Epub 2013 Sep 27. PMID 24077846
- [Derived] Mims AS, Kohlschmidt J, Borate U, Blachly JS, Orwick S, Eisfeld AK, Papaioannou D, Nicolet D, Mromicronzek K, Stein E, Bhatnagar B, Stone RM, Kolitz JE, Wang ES, Powell BL, Burd A, Levine RL, Druker BJ, Bloomfield CD, Byrd JC. A precision medicine classification for treatment of acute myeloid leukemia in older patients. J Hematol Oncol. 2021 Jun 23;14(1):96. doi: 10.1186/s13045-021-01110-5. PMID 34162404

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 58 participants were recruited.
Pre-assignment Details: One participant was deemed ineligible and is excluded from all analyses per study design.
Groups:
- Entire Cohort: All participants treatment on this study, see the Detailed Description for treatment information.
- Patients With HLA-matched Sibling Donor in Course 5: Patients undergo courses I-IV as in Detailed Description. Beginning 3-10 days after completion of course IV, patients with an HLA-matched sibling donor undergo total body irradiation (TBI) 2-3 times daily on days -7 to -4. Patients receive etoposide IV over 4 hours on day -3. Patients then undergo PBSCT on day 0. Patients then receive graft-vs-host disease prophylaxis with tacrolimus IV continuously on days -1 to 56 (or IV continuously on days -1 to 14 and then PO or IV every 12 hours on days 15-56) followed by a taper. Patients also receive methotrexate IV on days 1, 3, and 6, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 4 and continuing until blood counts recover. Patients then undergo course VI as in Detailed Description.
- Patients Without HLA-matched Sibling Donors in Course V: Patients undergo courses I-IV as in Detailed Description. Beginning 3-10 days after completion of course IV, patients without an HLA-matched sibling donor receive etoposide IV continuously and cytarabine IV over 2 hours on days 1-4. Patients also receive G-CSF SC beginning on day 14 and continuing until PBSC collection is complete. Patients receive imatinib mesylate PO twice daily beginning after completion of PBSC collection and continuing until 3 days before PBSCT. Patients then undergo TBI 2-3 times daily on days -8 to -5. Patients receive etoposide IV over 4 hours on day -4 and cyclophosphamide IV over 2 hours on day -2. Patients undergo PBSCT on day 0. Patients receive G-CSF SC beginning on day 0 and continuing until blood counts recover. Patients then undergo course VI as in Detailed Description.
- Patients Who Did Not Undergo Transplant for Course V: Patients undergo courses I-IV as in Detailed Description. Beginning 3-10 days after completion of course IV, patients who are not candidates for PBSCT receive etoposide IV over 4 hours and cytarabine IV over 2 hours on days 1-4. Patients also receive G-CSF SC once or twice a day beginning on day 14 and continuing until blood counts recover. Patients then undergo course VI as in Detailed Description.
Period: Initial Registration
Arm/Group | Entire Cohort | Patients With HLA-matched Sibling Donor in Course 5 | Patients Without HLA-matched Sibling Donors in Course V | Patients Who Did Not Undergo Transplant for Course V
Started | 57 | 0 | 0 | 0
Completed | 35 | 0 | 0 | 0
Not Completed | 22 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Relapsed | 6 | 0 | 0 | 0
Not completed — Received non-protocol therapy | 11 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0 | 0
Period: Course 5 (Transplant Assignments)
Arm/Group | Entire Cohort | Patients With HLA-matched Sibling Donor in Course 5 | Patients Without HLA-matched Sibling Donors in Course V | Patients Who Did Not Undergo Transplant for Course V
Started | 0 (After Course I-IV, participants were grouped into autologous, allogeneic or no transplant arms.) | 15 | 19 | 1
Completed | 0 | 15 | 19 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Cohort
Number analyzed (Participants) | 57
Age, Continuous [Median (Full Range); unit: years] | 44 [25 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 25
Region of Enrollment [Number; unit: participants]
  United States | 57

OUTCOME MEASURES:

1. Secondary Outcome: Overall Survival
Description: Overall survival (OS) as the interval from the on-study date until death. OS was estimated using the Kaplan Meier method.
Time Frame: Duration of study (up to 10 years)
Population: OS Analysis was powered to include all participants.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Entire Cohort
Number analyzed (Participants) | 57
years | 3.6 [1.9 to 6.2]

2. Secondary Outcome: Number of Participants Who Achieved a BCR-ABL Response at 12 Months
Description: BCR-ABL response is defined in two ways: complete molecular response (CMR) and major molecular response (MMR).
  Complete Molecular Response is defined as a Bcr-Abl (a fusion of gene of Bcr and ABl genes) ratio ≤0.0032% on the International Scale Bcr = breakpoint cluster gene Abl = abelson proto-oncogene
  MMR is defined as Bcr-Abl (A fusion gene of the breakpoint cluster region [Bcr] gene and Abelson proto-oncogene [Abl] genes) transcript ratio ≤0.1% (≥ 3 log reduction of BCR-ABL transcripts from a standardized baseline), as detected by reverse transcriptase polymerase chain reaction [RT-PCR] (performed centrally).
Time Frame: 12 months
Population: Peripheral blood stem cells were assayed from 13 patients.
Measure: Number; unit: participants
Arm/Group | Entire Cohort
Number analyzed (Participants) | 13
participants
  Complete Molecular Response | 9
  Major Molecular Response | 4

3. Primary Outcome: Disease Free Survival
Description: Disease-free survival (DFS) was measured as the interval from achievement of complete remission (CR) until relapse or death, regardless of cause; patients alive and in CR were censored at last follow-up. DFS was estimated using the Kaplan Meier method.
  A complete remission (CR) was defined as recovery of morphologically normal bone marrow and blood counts (i.e., neutrophils >= 1.5 x 10^9/L and platelets > 100 x 10^9/L) and no circulating leukemic blasts or evidence of extramedullary leukemia and persisting for at least one month.
Time Frame: Duration of treatment (up to 10 years)
Population: One participant was excluded per study design as they did not achieve a complete remission. DFS Analysis was powered to include all patients.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Entire Cohort
Number analyzed (Participants) | 56
years | 1.7 [1.1 to 4.1]

4. Secondary Outcome: 5 Year Disease-free Survival for Autologous & Allogeneic Transplant Groups
Description: Percentage of patients who achieved a complete remission (CR) and were alive and relapse free at 5 years. The 5-year progression free survival was estimated using the Kaplan Meier method.
Time Frame: 5 years from CR
Population: Participants who received autologous or allogeneic transplants were analyzed (N=34)
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Patients With HLA-matched Sibling Donor: Patients undergo courses I-IV as in Detailed Description. Beginning 3-10 days after completion of course IV, patients with an HLA-matched sibling donor undergo total body irradiation (TBI) 2-3 times daily on days -7 to -4. Patients receive etoposide IV over 4 hours on day -3. Patients then undergo PBSCT on day 0. Patients then receive graft-vs-host disease prophylaxis with tacrolimus IV continuously on days -1 to 56 (or IV continuously on days -1 to 14 and then PO or IV every 12 hours on days 15-56) followed by a taper. Patients also receive methotrexate IV on days 1, 3, and 6, and filgrastim (G-CSF) subcutaneously (SC) beginning on day 4 and continuing until blood counts recover. Patients then undergo course VI as in Detailed Description.
- Patients Without HLA-matched Sibling Donors: Patients undergo courses I-IV as in Detailed Description. Beginning 3-10 days after completion of course IV, patients without an HLA-matched sibling donor receive etoposide IV continuously and cytarabine IV over 2 hours on days 1-4. Patients also receive G-CSF SC beginning on day 14 and continuing until PBSC collection is complete. Patients receive imatinib mesylate PO twice daily beginning after completion of PBSC collection and continuing until 3 days before PBSCT. Patients then undergo TBI 2-3 times daily on days -8 to -5. Patients receive etoposide IV over 4 hours on day -4 and cyclophosphamide IV over 2 hours on day -2. Patients undergo PBSCT on day 0. Patients receive G-CSF SC beginning on day 0 and continuing until blood counts recover. Patients then undergo course VI as in Detailed Description.
Arm/Group | Patients With HLA-matched Sibling Donor | Patients Without HLA-matched Sibling Donors
Number analyzed (Participants) | 15 | 19
percentage of patients | 46 [26 to 80] | 47 [29 to 76]

5. Secondary Outcome: 5 Year Overall Survival for Autologous & Allogeneic Transplant Groups
Description: Percentage of patients who were alive at 5 years. The 5-year progression free survival was estimated using the Kaplan Meier method.
Time Frame: 5 years from registration
Population: Participants who were on autologous or allogeneic transplant arms were analyzed (N=34).
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Patients With HLA-matched Sibling Donor | Patients Without HLA-matched Sibling Donors
Number analyzed (Participants) | 15 | 19
percentage of patients | 53 [32 to 86] | 51 [32 to 80]

ADVERSE EVENTS:
Groups:
- Patients Who Did Not Undergo Transplant: Patients undergo courses I-IV as in Detailed Description. Beginning 3-10 days after completion of course IV, patients who are not candidates for PBSCT receive etoposide IV over 4 hours and cytarabine IV over 2 hours on days 1-4. Patients also receive G-CSF SC once or twice a day beginning on day 14 and continuing until blood counts recover. Patients then undergo course VI as in Detailed Description.
Arm/Group | Patients With HLA-matched Sibling Donor | Patients Without HLA-matched Sibling Donors | Patients Who Did Not Undergo Transplant
Serious Adverse Events (participants affected / at risk) | 6/15 | 9/19 | 3/23
Other Adverse Events (participants affected / at risk) | 15/15 | 19/19 | 21/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With HLA-matched Sibling Donor (N=15) | Patients Without HLA-matched Sibling Donors (N=19) | Patients Who Did Not Undergo Transplant (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 2 (3) | 0 (0)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (8) | 8 (10) | 3 (5)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2)
Edema (Cardiac disorders) | 2 (3) | 2 (2) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 2 (2) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 2 (2) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (2) | 0 (0) | 0 (0)
Dry eye syndrome (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorder (Eye disorders) | 2 (3) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis due to radiation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 2 (3) | 4 (5) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (8) | 7 (8) | 3 (4)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 6 (6) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (5) | 7 (7) | 2 (2)
Fever (General disorders) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 1 (1) | 4 (4) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 2 (2) | 5 (5) | 0 (0)
Infection without neutropenia (Infections and infestations) | 2 (2) | 3 (3) | 3 (3)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (6) | 7 (7) | 1 (2)
Alkaline phosphatase (Investigations) | 0 (0) | 1 (1) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (2) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 4 (6) | 5 (5) | 1 (2)
Blood bilirubin increased (Investigations) | 2 (2) | 3 (3) | 0 (0)
Creatinine increased (Investigations) | 3 (5) | 2 (3) | 0 (0)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
INR increased (Investigations) | 2 (3) | 1 (1) | 0 (0)
Leukocyte count decreased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 4 (5) | 7 (8) | 2 (3)
Platelet count decreased (Investigations) | 5 (9) | 8 (10) | 1 (2)
Weight loss (Investigations) | 2 (3) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 1 (1)
Blood glucose increased (Metabolism and nutrition disorders) | 5 (8) | 4 (4) | 2 (4)
Blood uric acid increased (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 1 (1)
Serum calcium decreased (Metabolism and nutrition disorders) | 4 (6) | 3 (3) | 2 (2)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Serum glucose decreased (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 0 (0)
Serum potassium decreased (Metabolism and nutrition disorders) | 3 (4) | 3 (4) | 2 (3)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 2 (3) | 2 (2) | 1 (1)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (2) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (painful urination) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urogenital disorder (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 3 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 4 (4) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1) | 3 (3) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With HLA-matched Sibling Donor (N=15) | Patients Without HLA-matched Sibling Donors (N=19) | Patients Who Did Not Undergo Transplant (N=23)
Blood disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 10 (10) | 1 (1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 14 (70) | 19 (149) | 19 (53)
Lymphatic disorder (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Transfusion: Platelets (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0)
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1 (2) | 2 (3) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 2 (3) | 0 (0)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac disorder (Cardiac disorders) | 1 (1) | 0 (0) | 1 (4)
Cardiac pain (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0)
Edema (Cardiac disorders) | 9 (24) | 10 (25) | 9 (13)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Myocardial ischemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Nodal arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 3 (4) | 3 (3) | 1 (1)
Sinus arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 4 (4) | 4 (11) | 0 (0)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ear disorder (Ear and labyrinth disorders) | 1 (3) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Cushingoid (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye syndrome (Eye disorders) | 3 (19) | 2 (2) | 0 (0)
Eye disorder (Eye disorders) | 3 (3) | 2 (2) | 1 (1)
Flashing vision (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 2 (3) | 1 (1) | 1 (1)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (4) | 6 (12) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (3) | 10 (14) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 12 (30) | 13 (42) | 9 (15)
Dry mouth (Gastrointestinal disorders) | 5 (13) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 4 (9) | 3 (3) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 4 (6) | 2 (3)
Gastrointestinal disorder (Gastrointestinal disorders) | 4 (7) | 3 (3) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Mucositis due to radiation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 14 (19) | 13 (16) | 2 (2)
Nausea (Gastrointestinal disorders) | 13 (39) | 18 (80) | 14 (28)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Stomatitis/pharyngitis (oral/pharyngeal mucositis) for BMT studies, if specified in (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 12 (23) | 15 (48) | 11 (17)
Chest pain (General disorders) | 0 (0) | 3 (5) | 1 (1)
Chills (General disorders) | 2 (5) | 6 (8) | 2 (2)
Edema limbs (General disorders) | 0 (0) | 4 (7) | 1 (2)
Fatigue (General disorders) | 11 (43) | 17 (77) | 12 (26)
Fever (General disorders) | 5 (5) | 6 (12) | 5 (6)
Ill-defined disorder (General disorders) | 1 (2) | 0 (0) | 0 (0)
Localized edema (General disorders) | 0 (0) | 1 (4) | 0 (0)
Pain (General disorders) | 4 (7) | 7 (19) | 5 (5)
Bladder infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gingival infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 4 (5) | 3 (4)
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 6 (8) | 8 (11) | 1 (1)
Infection without neutropenia (Infections and infestations) | 6 (10) | 11 (19) | 4 (5)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound-infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Postoperative hemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 4 (4) | 8 (13) | 0 (0)
Alanine aminotransferase increased (Investigations) | 10 (26) | 12 (36) | 7 (11)
Alkaline phosphatase (Investigations) | 4 (6) | 4 (6) | 2 (3)
Alkaline phosphatase increased (Investigations) | 1 (1) | 4 (4) | 4 (6)
Amylase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 11 (22) | 15 (44) | 9 (12)
Blood bilirubin increased (Investigations) | 6 (11) | 8 (11) | 2 (2)
Coagulopathy (Investigations) | 1 (1) | 0 (0) | 0 (0)
Creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Creatinine increased (Investigations) | 7 (14) | 8 (35) | 4 (5)
Electrocardiogram QTc interval prolonged (Investigations) | 0 (0) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (4) | 0 (0) | 0 (0)
INR increased (Investigations) | 3 (3) | 3 (5) | 1 (2)
Laboratory test abnormal (Investigations) | 1 (1) | 0 (0) | 2 (2)
Leukocyte count decreased (Investigations) | 7 (26) | 4 (28) | 9 (14)
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (8) | 3 (16) | 8 (14)
Neutrophil count decreased (Investigations) | 13 (42) | 17 (72) | 7 (20)
Platelet count decreased (Investigations) | 12 (43) | 19 (97) | 9 (14)
Weight gain (Investigations) | 5 (5) | 1 (3) | 1 (1)
Weight loss (Investigations) | 3 (3) | 2 (2) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 9 (15) | 13 (27) | 5 (5)
Blood glucose increased (Metabolism and nutrition disorders) | 9 (40) | 16 (62) | 12 (22)
Blood uric acid increased (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 2 (3) | 0 (0)
Serum albumin decreased (Metabolism and nutrition disorders) | 5 (9) | 8 (20) | 5 (8)
Serum calcium decreased (Metabolism and nutrition disorders) | 8 (20) | 10 (23) | 9 (12)
Serum glucose decreased (Metabolism and nutrition disorders) | 2 (2) | 6 (9) | 0 (0)
Serum magnesium decreased (Metabolism and nutrition disorders) | 8 (16) | 8 (16) | 1 (1)
Serum magnesium increased (Metabolism and nutrition disorders) | 1 (1) | 3 (3) | 0 (0)
Serum phosphate decreased (Metabolism and nutrition disorders) | 4 (9) | 6 (9) | 3 (3)
Serum potassium decreased (Metabolism and nutrition disorders) | 8 (17) | 14 (49) | 9 (14)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (2) | 3 (4) | 0 (0)
Serum sodium decreased (Metabolism and nutrition disorders) | 4 (11) | 5 (10) | 4 (5)
Serum sodium increased (Metabolism and nutrition disorders) | 1 (2) | 1 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7) | 6 (9) | 3 (6)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (5) | 0 (0) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Joint disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (6) | 3 (3) | 1 (1)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (13) | 10 (23) | 5 (9)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (5) | 0 (0)
Arachnoiditis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 2 (3) | 0 (0)
Dizziness (Nervous system disorders) | 5 (10) | 9 (14) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (7) | 1 (1) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 12 (28) | 17 (40) | 12 (14)
Memory impairment (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
Neurological disorder NOS (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0)
Nystagmus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 4 (4) | 5 (12) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 9 (20) | 14 (48) | 10 (17)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 8 (15) | 2 (3) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (7) | 7 (11) | 3 (3)
Confusion (Psychiatric disorders) | 5 (5) | 4 (4) | 2 (2)
Depression (Psychiatric disorders) | 3 (6) | 7 (11) | 3 (4)
Insomnia (Psychiatric disorders) | 4 (4) | 7 (10) | 3 (4)
Dysuria (painful urination) (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Hematuria (in the absence of vaginal bleeding) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage urinary tract (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
Urine discoloration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urogenital disorder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Gynecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Reproductive tract disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Testicular pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (10) | 3 (4)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (16) | 12 (23) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (3) | 0 (0)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 9 (12) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 6 (10) | 5 (9) | 3 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (4) | 3 (3) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hand-and-foot syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 0 (0)
Photosensitivity (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (2) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (4) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Rash desquamating (Skin and subcutaneous tissue disorders) | 11 (20) | 11 (16) | 5 (6)
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash/desquamation associated with graft versus host disease (GVHD) for BMT studies (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (3) | 0 (0)
Sweating (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Flushing (Vascular disorders) | 2 (2) | 1 (1) | 0 (0)
Hemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 2 (2) | 2 (2) | 0 (0)
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 2 (2) | 0 (0) | 0 (0)
Hot flashes (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (5) | 4 (6) | 2 (2)
Hypotension (Vascular disorders) | 2 (2) | 3 (6) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1) | 3 (5) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less